CLINICAL TRIAL: NCT06512987
Title: Effects of Technology-Driven, Interactive Intensive Care Unit Diary on Psychological Distress in Patients Requiring Intensive Care: A Randomized Controlled Trial
Brief Title: Impact of Interactive ICU Diary on Psychological Distress
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to insufficient staffing, which impacted the ability to continue subject enrollment and study operations.
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N202403088
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-07

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interactive ICU Diary Group (Experimental): Patients in this group will use a technology-driven, interactive ICU diary from the first day of ICU admission until discharge. Through the diary platform, patients can share their feelings and needs, while family members can send supportive messages, pictures, and videos. Healthcare providers will use the platform to connect with families and monitor patient conditions. The goal is to reduce psychological distress, specifically anxiety, depression, and stress, during the ICU stay.
  Interventions: Other: technology-driven, interactive ICU diary
- routine care (No Intervention): Patients in this group will receive standard ICU care without the use of the interactive ICU diary.

INTERVENTIONS:
Other: technology-driven, interactive ICU diary — Through the diary platform, patients can share their feelings and needs, while family members can send supportive messages, pictures, and videos. Healthcare providers will use the platform to connect with families and monitor patient conditions.
  Arms: Interactive ICU Diary Group

SUMMARY:
This study investigates the effectiveness of a technology-driven, interactive ICU diary in reducing psychological distress, specifically anxiety, depression, and stress, in ICU patients. A single-blind, parallel-group randomized controlled trial will include 56 conscious ICU patients. The primary outcome measures are the Depression, Anxiety, and Stress Scale-21 (DASS-21) and the EuroQol instrument (EQ-5D), assessed at ICU admission, discharge, and one month post-discharge.

DETAILED DESCRIPTION:
This study investigates the effectiveness of a technology-driven, interactive ICU diary in reducing psychological distress, specifically anxiety, depression, and stress, in ICU patients. A single-blind, parallel-group randomized controlled trial will include 56 conscious ICU patients, randomly assigned to either the interactive diary group or the standard care group. The interactive diary allows patients to share their feelings and needs via a platform, while family members can send supportive messages, pictures, and videos. Healthcare providers can connect with families and monitor patient conditions through the platform. The primary outcome measures are the Depression, Anxiety, and Stress Scale-21 (DASS-21) and the EuroQol instrument (EQ-5D), assessed at ICU admission, discharge, and one month post-discharge. The expected results indicate that the interactive diary will significantly alleviate psychological distress during the ICU stay and improve post-discharge quality of life, providing valuable insights into enhancing the mental health and overall well-being of ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clear consciousness and able to communicate in Mandarin, Taiwanese, or Hakka
* Expected ICU stay of at least 72 hours
* Ability to operate a smart device and use social media applications

Exclusion Criteria:

* Presence of delirium before joining the study (Intensive Care Delirium Screening Checklist score ≥ 4)
* Physical, auditory, or visual impairments preventing the use of smart devices History of epilepsy, cognitive impairments (e.g., hepatic encephalopathy, dementia), or psychiatric disorders
* Richmond Agitation-Sedation Scale score not between +1 and -1 (indicating excessive sedation or agitation)
* Acute Physiology and Chronic Health Evaluation Score (APACHE-II) > 25 within the first 24 hours of ICU admission (indicating > 50% mortality rate)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Psychological Distress Levels (DASS-21) | 7 days after admission and one month post-discharge.
  The primary outcome will be the psychological distress levels measured by the Depression, Anxiety, and Stress Scale-21 (DASS-21). This scale assesses anxiety, depression, and stress in ICU patients through 21 items, each rated from 0 ("Did not apply to me at all - Never") to 3 ("Applied to me very much, or most of the time - Almost always"). The total score for each subscale (DASS-21-Depression, DASS-21-Anxiety, and DASS-21-Stress) ranges from 0 to 21, with higher scores indicating greater emotional distress. The cutoff scores for DASS-21-Depression, DASS-21-Anxiety, and DASS-21-Stress are >9, >7, and >14, respectively.

SECONDARY OUTCOMES:
Quality of Life (EQ-5D) | 7 days after admission and one month post-discharge.
  The secondary outcome will be the quality of life measured by the EuroQol instrument (EQ-5D-3L). This instrument includes five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is scored with three levels: no problems (1), some problems (2), and extreme problems (3). The EQ-5D index score, derived using a pre-established conversion formula from neighboring countries like Japan or the UK, ranges from 0 to 1, with higher scores indicating better quality of life. Additionally, the EQ-VAS, a visual analogue scale from 0 (worst imaginable health) to 100 (best imaginable health), will be used to assess self-perceived health status. The EQ-VAS score will be recorded directly by marking a vertical scale.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yean Chiu, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No